CLINICAL TRIAL: NCT04833595
Title: Can Mindful Eating Improve Cholesterol and Glucose Level: A Tele-Health Pilot-Randomised Controlled Trial
Brief Title: Can Mindful Eating Improve Cholesterol and Glucose Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monash University Malaysia (Other)
Responsible Party: Principal Investigator, Teoh Siew Li, Lecturer, Monash University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27779
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cholesterol; Lipidosis
MeSH Terms: conditions — Lipidoses

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Arm (Experimental): A recommendation on healthy food intake will be sent to participants. At the end of each week, participants will be required 1) to submit THREE photos of the meals that they are most satisfied with in terms of healthiness and 2) using the photos to answer a questionnaire about their diet. The photos and completed questionnaire must be submitted to the research investigator each week for a total of 8 weeks. After 8 weeks, participants will be required to get tested for your fasting total cholesterol and blood glucose level in the appointed pharmacy for the second time. It is estimated to require 15-30 minutes of their time weekly.
  The questionnaire used for experimental group contains reflective questions as part of the mindfulness intervention.
  Interventions: Behavioral: Mindfulness practice
- Non-mindfulness Arm (Active Comparator): Everything is similar to the experimental arm. However, the questionnaire used for control group does not contain reflective questions to serve as control group.
  Interventions: Behavioral: Mindfulness practice

INTERVENTIONS:
Behavioral: Mindfulness practice — Mindfulness is hypothesised to include reflective practice. Therefore, reflective questions are asked in the questionnaire for intervention group but not for control group.

SUMMARY:
This study aims to explore the effectiveness of mindful eating and its effect on cholesterol and glucose level. The participants will be required to get tested for their fasting total cholesterol and blood glucose level for two times. At the first visit, they will be required to complete the survey given and be tested for their fasting total cholesterol and blood glucose level. A recommendation on healthy food intake will be sent to participants. At the end of each week, participants will be required 1) to submit THREE photos of the meals that they are most satisfied with in terms of healthiness and 2) using the photos to answer a questionnaire about their diet. The photos and completed questionnaire must be submitted to the research investigator each week for a total of 8 weeks. After 8 weeks, participants will be required to get tested for their fasting total cholesterol and blood glucose level in the appointed pharmacy for the second time. It is estimated to require 15-30 minutes of their time weekly.

DETAILED DESCRIPTION:
Consistently high cholesterol or/and glucose level pose harmful threat to the body that may cause lethal health conditions (e.g. stroke, cardiovascular diseases). In addition, 3.6 million Malaysians are suffering from diabetes, the highest rate of incidence in Asia and one of the highest in the world. There is crucial need to find ways to improve the situation. Tele-health interventions and mindful eating behaviours are proposed to be effective in improving the levels of cholesterol and glucose. To investigate and explore the intervention, a small-scale randomised controlled trial will be conducted by comparing the effectiveness of mindful eating and the effect on cholesterol and glucose level. Students will collect and analyse both quantitative and qualitative data.

A small-scale randomised controlled trial will be conducted to compare the effectiveness of mindful eating and the effect on lipid level. Subjects will be randomly assigned to intervention or control group. For intervention group, subjects will be required to snap picture of every meal that they consume. At the end of the day, they are required to actively recall and reflect on how healthy they consider their meals to be. The reflection will be submitted to the research team daily together with the taken pictures of meal. As for the control group, subjects will only snap and submit the picture of their meals but without active recall and reflection.

Subjects are required to return to the community pharmacy after two months to follow-up on their glucose and lipid levels post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Total fasting cholesterol of at least 5.2mmol/L

Exclusion Criteria:

* Familial hypercholesterolaemia or Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting total cholesterol | 8 weeks
  Total cholesterol taken after at least 8 hours fasting

SECONDARY OUTCOMES:
Fasting glucose | 8 weeks
  Blood glucose taken after at least 8 hours fasting

CONTACTS AND LOCATIONS:
Overall Officials: Phaik Eong Poh, PhD, Study Director — Monash University Malaysia
Locations (1):
- Monash University Malaysia, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be shared upon request to investigator.